CLINICAL TRIAL: NCT03714243
Title: A Study to Evaluate the Safety and Feasibility of Blood-Brain Barrier Disruption Using MRI-Guided Focused Ultrasound in the Treatment of Her2-positive Breast Cancer Brain Metastases
Brief Title: Blood Brain Barrier Disruption (BBBD) Using MRgFUS in the Treatment of Her2-positive Breast Cancer Brain Metastases
Acronym: BBBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BT006; 277990 (Other: Health Canada)
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer; Brain Metastases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, single center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ExAblate BBBD (Experimental): Using ExAblate Model 4000 Type-2 to temporarily disrupt the blood brain barrier in patients with Her-2 positive breast cancer and brain metastases
  Interventions: Device: ExAblate BBBD

INTERVENTIONS:
Device: ExAblate BBBD — Using ExAblate Model 4000 Type-2 to temporarily disrupt the blood brain barrier in patients with Her-2 positive breast cancer and brain metastases
  Other Names: Exablate Neuro

SUMMARY:
The purpose of this study is to evaluate the safety of BBB disruption using the ExAblate 4000-system Type 2 in patients with Her-2 positive breast cancer metastases in the brain.

DETAILED DESCRIPTION:
The goal of this prospective, single arm, non-randomized study is to evaluate the safety and feasibility of using the Exablate Model 4000 Type 2 "Neuro-System" as a tool to serially disrupt the blood brain barrier in a temporary and localized fashion in patients with breast cancer and brain metastases. Up to 10 patients will be recruited at Sunnybrook. Patients will be consented, screened, undergo up to 6 study Exablate BBBD treatment cycles, every 2-3 weeks based on their trastuzumab regimen. Follow-up will continue through 12 weeks following the last BBBD post-treatment and the subject's participation in the study will be complete.

Data will be collected to establish the basic safety of this type of treatment as the basis for later studies to evaluate clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 80 years of age
* Able and willing to give informed consent
* Metastatic Her2-positive breast cancer with brain metastases
* Karnofsky performance score 70-100
* ASA score 1-3
* Able to communicate sensations during the ExAblate BBBD procedure
* Able to attend all study visits (i.e., life expectancy of at least 3 months)
* At least 14 days passed since last brain surgery
* At least 6 weeks passed since last radiation treatment

Exclusion Criteria:

* Brain metastases not visible on the pre-therapy imaging
* The sonication pathway to the tumour involves:

  i. Extensive scalp scars ii. Clips or other metallic implanted objects in the skull or the brain, except shunts
* The subject presents with symptoms and signs of increased intracranial pressure (e.g., headache, nausea, vomiting, lethargy, and papilledema)
* Cardiac disease or unstable hemodynamics including:

  i. Documented myocardial infarction within six months of enrolment ii. Unstable angina on medication iii. Congestive heart failure iv. Left ventricular ejection fraction < 50% v. Right-to-left, bidirectional, or transient right-to-left cardiac shunts vi. History of a hemodynamically unstable cardiac arrythmia vii. Cardiac pacemaker viii. Contraindications to perflutren including subjects with a family or personal history of QT prolongation or taking concomitant medications known to cause QTc prolongation
* Severe hypertension (diastolic BP > 100 on medication)
* Anti-coagulant therapy or medications known to increase risk of hemorrhage within washout period prior to treatment (i.e. antiplatelet or vitamin K inhibitor anticoagulants within 7 days, non-vitamin K inhibitor anticoagulants within 72 hours, or heparin-derived compounds within 48 hours of treatment)
* History of a bleeding disorder, coagulopathy or with a history of spontaneous tumour hemorrhage
* Abnormal level of platelets (< 100000) or INR > 1.3
* Documented cerebral infarction within the past 12 months
* Transient Ischemic Attack (TIA) in the last 1 month
* Known allergy sensitivity or contraindications to gadolinium-diethylenetriamine penta-acetic acid (DTPA), CT contrast, or perflutren or trastuzumab
* Allergy to eggs or egg products
* Contraindications to MRI such as non-MRI-compatible implanted devices
* Large subjects not fitting comfortably into the MRI scanner (generally >250 lbs)
* Difficulty lying supine and still for up to 4 hours in the MRI unit or claustrophobia
* Untreated, uncontrolled sleep apnea
* Positive pregnancy test (for pre-menopausal women)
* Known life-threatening systemic disease
* Severely impaired renal function
* Respiratory: chronic pulmonary disorders, e.g. severe emphysema, chronic obstructive pulmonary disease (COPD), pulmonary vasculitis, or other causes of reduced pulmonary vascular cross-sectional area, subjects with a history of drug allergies
* Any illness or medical condition that in the investigator's opinion precludes participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Adverse events | Throughout the study, approximately 10 months.
  Rate of adverse events following each treatment through end of study

SECONDARY OUTCOMES:
Feasibility of BBBD | Immediately after each BBBD procedure
  The extent of BBB opening will be determined by the degree of contrast enhancement seen on post-procedure MRI with contrast agent

CONTACTS AND LOCATIONS:
Overall Officials: Nir Lipsman, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada